CLINICAL TRIAL: NCT06434857
Title: Effectiveness of a Strength Program Over Cognitive Functionality in Older Adults Undergoing an Occupational Therapy Program
Brief Title: Effectiveness of a Strength Program Over Cognitive Functionality in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Arturo Dávila Marcos, PhD student, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16069701
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Impairment; Aging Problems
Keywords: Aging; Cognitive impairment; Older adult; Strength training; Therapeutic exercise
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Resistance Training; Aging

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strength Training Group (Experimental): The main part of the strength training program will have the following exercises: wall push-ups, arm raises, elbow push-ups and extensions, weighted pronosupination, hand press, knee and hip hinge squat, deadlifts, front and sagittal plan stride, and heel raises.
  It will consist on different phases:
  1. st phase: exercise adaptation: the correct execution of upper and lower limb exercises will be taught for one month.
  2. nd phase: Resistance training: During the following seven months, strength exercises will be performed at slow and normal speed of the movement patterns learned in the training course, increasing load and volume according to each subject's individual progress.
  Interventions: Procedure: Strength training in older adults with mild or non existent cognitive impairment
- Multimodal Exercise Group (Active Comparator): The main part of the multicomponent exercise program integrates different exercise modalities: Aerobic, mobility, strength, balance and coordination exercises. Playful activities or games are also included.
  Exercises will be turned gradually more demanding along the duration of the program.
  Interventions: Procedure: Multimodal excercise in older adults with mild or non existent cognitive impairment
- Control Group (No Intervention): Participants in this group should continue with their usual dietary pattern and level of physical activity, without changing their lifestyle habits during the study period. They will not participate in the strength exercise program, nor will they perform systematic, programmed and supervised physical exercise in any other program.

INTERVENTIONS:
Procedure: Strength training in older adults with mild or non existent cognitive impairment — Strength training program applied to strength training group
  Arms: Strength Training Group
Procedure: Multimodal excercise in older adults with mild or non existent cognitive impairment — Multimodal exercise program applied to multimodal exercise group
  Arms: Multimodal Exercise Group

SUMMARY:
This is a randomized, parallel, double-blind clinical trial. The main objective is to compare the efficacy of strength training, multimodal exercise with non-specific exercises and a control group on cognitive functionality and physical composition in subjects over 65 years of age with mild or non existent cognitive impairment currently receiving occupational therapy.

The intervention in both groups will be carried out for 30 weeks, with three weekly sessions. Two evaluations will be performed, one pre-intervention and one post-intervention. Cognitive Functionality (Montreal Cognitive Assessment (MOCA) and Lawton and Brody Scale), Sleep quality (Athens insomnia scale and Pittsburgh sleep quality index), physical functionality (Timed up and go (TUG), chair stand test and hand grip test and Short Physical Performance Battery (SPPB)), body composition (Body fat %, skeletal muscle index (SMI), appendicular skeletal muscle (ASM), waist circumference, waist hip ratio, body weight, body mass index (BMI)) will be evaluated.

DETAILED DESCRIPTION:
Design: Randomized, controlled clinical trial with three parallel groups, in which subjects over 65 years of age will be recruited. Study participants will be assigned to one of the three intervention groups. The study will have a duration of 8 months. There will be 2 evaluation visits, an initial one, and a final one after 8 months. During 8 months there will be 3 weekly sessions lasting 50 minutes.

Scope: The study will be carried out in the Salamanca Health Area, in collaboration with the Research, Teaching and Assistance Unit of the Faculty of Nursing and Physiotherapy of the University of Salamanca and the Department of Elderly People of the Salamanca City Council.

Interventions: 1) Multimodal Exercise Group (GEM); 2) Strength Exercise Group (GES); 3) No Exercise Control Group (CG). The GEM and GES sessions follow the same structural pattern. They will be structured according to the recommendations of the American College of Sports Medicine (ACSM). In the main part of the GES, only strength exercises will be performed.

Study population: 90 subjects over 65 years of age from the city of Salamanca will be recruited, distributed in 3 groups at a 1:1:1 ratio. Randomization will be performed using the Epidat 4.2 program. The sample size was calculated using GRANMO Version 7. 12 April 2012.

The main study variables are: Cognitive functionality (Montreal Cognitive Assessment (MOCA) and Lawton and Brody Scale), Sleep quality (Athens insomnia scale and Pittsburgh sleep quality index), Physical Functionality (Timed Up & Go test (TUG), chair stand test and hand grip test and Short Physical Performance Battery (SPPB)), body composition (Body fat %, skeletal muscle index (SMI), appendicular skeletal muscle (ASM), waist circumference, waist hip ratio, body weight, body mass index (BMI)), SARC-F Questionnaire, % RM estimated by force-velocity profile and Gait speed.

Population characteristics will be presented as mean and standard deviation for continuous variables and as frequency distribution for qualitative variables. Statistical analysis The effect of the intervention on the study variables if the variables are parametric, Student's t-test will be used, and if they are non-parametric, the Wilcoxon test will be used. An alpha risk of 0.05 is set as the limit of statistical significance. The statistical program to be used will be SPSS, v.26.0.

The study will be carried out with the authorization of the Ethics Committee on Drug Research (CEIm) of the Salamanca Health Area, and with the prior informed consent of the study subjects. The participants will be informed of the objectives of the project and of the risks and benefits of the examinations and interventions to be performed. The study has been designed and subsequently assessed in accordance with Law 14/2007 on Biomedical Research, the ethical principles of the Declaration of Helsinki of the World Medical Association on ethical principles for medical research involving human subjects, as well as the other ethical principles and legal regulations applicable according to the characteristics of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 65

Exclusion Criteria:

* Absolute contraindication for excersice
* Severe cognitive impairment or dementia
* Language barriers
* Pending litigation or legal claim

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Cognitive functionality | 8 months
  Cognitive functionality will be measured with the Montreal Scales Assessment (MOCA). Maximum score is 30, considering a punctuation ≥ 26 is considered normal.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | 6 months
  A questionaire consisting of 7 items to screen sleep quality: subjective sleep quality,sleep latency, sleep duration, usual sleep efficiency, sleep perturbations, use of medication and daytime disfunction. Each item is scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Athens insomnia scale | 6 months
  A shorter and simpler questionaire to quickly screen sleep quality. It consists of 8 components, each one scored from 0 to 3. Higher scores indicate worse sleep quality.
Body Mass Index (BMI) | 8 months
  It is a measure used to assess a person's body weight in relation to their height. It is calculated by dividing a person's weight in kilograms by their height in meters squared (BMI = kg/m²).
Short Physical Performance Battery (SPPB) | 8 months
  Test battery to assess physical performance and frailty degree consisting of 3 tests: gait speed, balance, and lower limb strength. The maximum score is 12 points and a score ≤ 8 points indicates poor physical performance.
Gait speed | 8 months
  It is considered a fast, safe and very reliable test for sarcopenia, in a distance of 4 meters, values greater than 0.8 m/s are considered positive.
Timed Up and Go (TUG) | 8 months
  A predictive test for frailty and falls, where individuals are asked to get up from a standard chair, walk to a marker 3 m away, turn around, and sit down again. Times greater than 20 seconds are considered positive.
Lawton & Brody Scale | 8 months
  A scale to evaluate functionality and independence in daily activities. It screens 8 items, ranged from 0 to 1. For women, a score of 8 is considered autonomous while for men the score is 5.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Dávila Marcos, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No